CLINICAL TRIAL: NCT00528164
Title: Treating Childhood Obesity With Family Lifestyle Change
Brief Title: Team PLAY (Positive Lifestyles for Active Youngsters)
Acronym: Team PLAY
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1RO1HDO50895-01; USPHS Gr HD-050895-01
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Obesity
Keywords: children; overweight; obesity; family; intervention; control; randomized; physical activity; diet; nutrition; behavior; body mass index
MeSH Terms: conditions — Obesity; Overweight; Motor Activity; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Team PLAY Group (Experimental): 6-month family-centered intervention to increase physical activity and healthy eating patterns, primarily directed at parents. Parents will receive intense counseling regarding developmentally appropriate physical activity, strategies for reducing sedentary behaviors, nutritional counseling, and behavioral counseling, including a self-management program to use with their children at home. The group will meet once a week for the initial 8 weeks, bi-weekly for 8 weeks, and monthly for 2 months.
  Interventions: Behavioral: Team PLAY
- Standard Care Group (No Intervention): Participants receive standard care by primary care physician.

INTERVENTIONS:
Behavioral: Team PLAY — Parents will receive intense counseling regarding developmentally appropriate physical activity, strategies for reducing sedentary behaviors, nutritional counseling, and behavioral counseling, including a self-management program to use with their children at home. The group will meet once a week for the initial 8 weeks, bi-weekly for 8 weeks, and monthly for 2 months.
  Arms: Team PLAY Group

SUMMARY:
The purpose of this study is to determine whether an intense family-centered program to help children, 4 to 7 years old, control their weight is more effective than the advise and referrals their health provider gives in the primary care office.

DETAILED DESCRIPTION:
This randomized controlled trial is designed to determine whether an intense 6 month family-centered intervention to increase physical activity and health eating patterns, primarily directed at parents, followed by a 6 month maintenance period, will be significantly more successful in controlling weight in overweight/obese children, ages 4-7 years, than usual standard care, at 2 years after enrollment. The intervention group (180 children with a BMI > 85% percentile) will receive standard of care, as well as, additional parental counseling. Parents will receive intense counseling regarding developmentally appropriate physical activity, strategies for reducing sedentary behaviors, nutritional counseling, and behavioral counseling including a self-management program to use with their children at home. The group will meet once a week for the initial 8 weeks, biweekly for 8 weeks, and monthly for 2 months. Following this period (the next 6 months), a case manager will call the family on a monthly basis and the family will be sent educational and support information by mail. The control group (60 children with a BMI > 85% percentile) will receive standard care provided by their primary care provider and be offered a six week optional parenting class. All children will have a medical history, physical examination, and anthropometric measures, nutritional assessment, measurement of physical activity, and behavioral/psycho-social measures provided by study personnel. Outcome measurements will be done at baseline, 6, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Children 4 to 7 years of age, male or female, of any race who have a BMI > 85% for age.
* All participants and parents must be able to speak and understand English.

Exclusion Criteria:

* History of diabetes mellitus
* History of significant renal, hepatic, cardiovascular,or gastrointestinal disease
* Receiving drugs known to alter glucose homeostasis
* Physical disabilities that limit physical activity (i.e. orthopedic, congenital)
* Diagnosis of hypertension by a medical provider that requires limited physical activity
* Psychological disabilities that might limit participation;
* Lack of access to a telephone
* Lack of access to transportation for the intervention
* Current participation in another clinical trial (current participation in an observational study is not an exclusion.)
* Other medical or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol.
* Unable to speak and understand English

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 270 (Actual)
Dates: Start 2006-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Primary - Body Mass index | 2 years

SECONDARY OUTCOMES:
Body Composition (DXA), physical activity (accelerometry), dietary changes (Block Food Frequency), Flexibility and Cohesion Evaluation Scales, MacArthur Behavior and Health Questionnaire and Body Esteem Scale. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marion E Hare, MD,MS, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee, Department of Preventive Medicine, Memphis, Tennessee, United States

REFERENCES:
- [Background] Williams NA, Fournier J, Coday M, Richey PA, Tylavsky FA, Hare ME. Body esteem, peer difficulties and perceptions of physical health in overweight and obese urban children aged 5 to 7 years. Child Care Health Dev. 2013 Nov;39(6):825-34. doi: 10.1111/j.1365-2214.2012.01401.x. Epub 2012 Aug 8. PMID 22882115
- [Background] Hare ME, Coday M, Williams NA, Richey PA, Tylavsky FA, Bush AJ. Methods and baseline characteristics of a randomized trial treating early childhood obesity: the Positive Lifestyles for Active Youngsters (Team PLAY) trial. Contemp Clin Trials. 2012 May;33(3):534-49. doi: 10.1016/j.cct.2012.02.003. Epub 2012 Feb 10. PMID 22342450
- [Background] Williams NA, Coday M, Somes G, Tylavsky FA, Richey PA, Hare M. Risk factors for poor attendance in a family-based pediatric obesity intervention program for young children. J Dev Behav Pediatr. 2010 Nov-Dec;31(9):705-12. doi: 10.1097/DBP.0b013e3181f17b1c. PMID 21057255